CLINICAL TRIAL: NCT06125964
Title: Using Real-Time Data Capture to Examine Affective Mechanisms as Mediators of Physical Activity Adherence in Interventions: Formative Study
Brief Title: eMOTION Formative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Genevieve Dunton, Chief, Division of Health Behavior Research and Director, USC Real-Time Eating Activity and Children's Health (REACH) Lab, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: UP-22-00332-formative; R01CA272933 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Physical Inactivity; Overweight or Obesity; Cancer
Keywords: Affective Response; Psychological Needs; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity; Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Treatment components targeting intensity-based goals and affect-based goals will be tested separately in four groups of n=9 participants: (1) intensity-based goal setting alone; (2) affect-based goals + TYPE/CONTEXT; (3) affect-based goals + SAVOR; and (4) affect-based goals + TYPE/CONTEXT + SAVOR.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The majority of study staff will be blinded to participant assignment for most of the study period. Data will be analyzed blind to allocation, and participants will be blind to their allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intensity (Experimental): Participants receive intensity-based goals for two weeks. No enhancements are added to the standard mHealth intervention.
  Interventions: Behavioral: Intensity-Based Goals
- Affect + TYPE/CONTEXT (Active Comparator): Participants receive affect-based goals for two weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT enhancement to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Affect-Based Goals; Behavioral: TYPE/CONTEXT Enhancement
- Affect + SAVOR (Active Comparator): Participants receive affect-based goals for two weeks. In addition to the standard mHealth intervention, participants engage in the SAVOR enhancement to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Affect-Based Goals; Behavioral: SAVOR Enhancement
- Affect + TYPE/CONTEXT + SAVOR (Active Comparator): Participants receive affect-based goals for two weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT and SAVOR enhancements to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Affect-Based Goals; Behavioral: TYPE/CONTEXT Enhancement; Behavioral: SAVOR Enhancement

INTERVENTIONS:
Behavioral: Intensity-Based Goals — On days participants plan to exercise, morning and evening goal sessions ask them to provide an activity goal for the day; create a concrete plan; prompt them to anticipate barriers and brainstorm solutions; and reflect on whether they were able to meet this goal. Intensity-based goals ask participants to maintain a target heart rate range during physical activity based on age-adjusted heart rate (HR) max. Goals progressively increase from 55% to 60% HR max across two weeks. Research staff will show participants how to monitor their heart rate using their Fitbit Versa. For each condition, the Fitbit Versa device will feature a custom watch face with a clock (current local time), the date, current device battery levels, and an exercise button. The exercise button can be pressed whenever a subject wants to engage in physical activity, and provides real-time feedback on heart rate (intensity-based goals only) and exercise duration.
  Arms: Intensity
Behavioral: Affect-Based Goals — On days participants plan to exercise, morning and evening goal sessions ask them to provide an activity goal for the day; create a concrete plan; prompt them to anticipate barriers and brainstorm solutions; and reflect on whether they were able to meet this goal. Affect-based goals ask participants to engage in either a type or context of physical activity that allows them to experience positive affect. Goals focused on context are randomly generated to suggest that the participant performs activity in a place, in a social situation, or while listening to something that makes them feel good. For each condition, the Fitbit Versa device will feature a custom watch face with a clock (current local time), the date, current device battery levels, and an exercise button. The exercise button can be pressed whenever a subject wants to engage in physical activity, and provides real-time feedback on exercise duration while featuring a "smiley face" emoticon.
  Arms: Affect + SAVOR; Affect + TYPE/CONTEXT; Affect + TYPE/CONTEXT + SAVOR
Behavioral: TYPE/CONTEXT Enhancement — The TYPE/CONTEXT enhancement will augment affect-based treatment effects by additionally providing tailored recommendations for activity types and contexts that satisfy personally important psychological needs as rated by each participant at baseline. Ratings from a crowdsourced panel of adults on Amazon Mechanical Turk were used to determine the potential for specific activity types and contexts to satisfy psychological needs; our tailoring algorithm recommends the corresponding activity type or context while accounting for reported constraints. Different psychological needs will be selected each day. Tailored recommendations are incorporated immediately following the morning goal module.
  Arms: Affect + TYPE/CONTEXT; Affect + TYPE/CONTEXT + SAVOR
Behavioral: SAVOR Enhancement — The SAVOR enhancement will augment affect-based treatment effects by additionally implementing a brief savoring exercise on the smartphone during the evening goal session (after the self-monitoring module). Participants will respond to questions that are intended to enhance and prolong positive experiences during physical activity. To trigger attentional deployment, a common savoring strategy that involves intensifying experiences by focusing on them, participants will answer open-ended prompts. These prompts are drawn from a prompt pool with slightly varied wording to promote a sense of novelty.
  Arms: Affect + SAVOR; Affect + TYPE/CONTEXT + SAVOR

SUMMARY:
The eMOTION Study is a two-part ORBIT model phase 1 trial. The first part, called the Formative Study, will assess acceptability and feasibility of a novel physical activity intervention in adults at increased risk for cancer due to overweight or obesity.

DETAILED DESCRIPTION:
The eMOTION Study is a two-part ORBIT model phase 1 trial. The first part of the eMOTION Study, the Formative Study, will iteratively test and refine the implementation of a novel treatment to manipulate affective mechanisms during physical activity among individuals at higher risk for cancer due to overweight or obesity. Acceptability and feasibility of content, delivery, device usage, engagement, and achieving clinically meaningful changes in affective mechanisms will be addressed. Treatment components targeting intensity-based goals and affect-based goals will be tested separately in four groups.

ELIGIBILITY:
Inclusion Criteria:

* adults aged ≥18 years
* residing in the United States
* self-reported BMI ≥ 25
* currently engaging in < 60 minutes per week of structured physical activity
* owning a personal smartphone device
* residing in an area with Internet or Wi-Fi connectivity during the study period
* able to speak and read in English
* interested and willing to start a physical activity program
* willing to wear a Fitbit Versa smartwatch provided by the study team everyday continuously (including at work and during physical activity), in place of any Fitbits or smartwatches they previously wore, for the duration of the study period
* able to read the small font on a smartwatch screen without glasses, or willing to carry reading glasses during physical activity for the purpose of reading the smartwatch screen

Exclusion Criteria:

* unable to provide informed consent due to cognitive disability
* unable to engage in one or more key treatment components, including those with medical conditions that preclude physical activity engagement or who cannot wear an accelerometer on the wrist for any reason
* currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve F Dunton, PhD MPH, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment, onboarding continued with a baseline questionnaire, a Fitbit smartwatch sent in the mail, and orientation session attendance. Then, a week-long run-in period allowed for assessment components (e.g., Fitbit smartwatch monitoring, check-ins) to be gradually introduced. n=9 participants were lost due to technological issues experienced during onboarding and the run-in period, so N=37 participants were randomly assigned to groups.
Groups:
- Affect + TYPE/CONTEXT: Participants receive affect-based goals for two weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT enhancement to augment the treatment effects of the affect-based goals condition.
  Affect-Based Goals: On days participants plan to exercise, they engage in affect-based goal-setting sessions. Participants are asked to engage in a type or context of physical activity that allows them to experience positive affect.
  TYPE/CONTEXT Enhancement: The TYPE/CONTEXT enhancement will augment affect-based treatment effects by additionally providing tailored recommendations for activity types and contexts that satisfy personally important psychological needs as rated by each participant at baseline. Ratings from a crowdsourced panel of adults on Amazon Mechanical Turk were used to determine the potential for specific activity types and contexts to satisfy psychological needs; our tailoring algorithm recommends the corresponding activity type or context while accounting for reported constraints. Different psychological needs will be selected each day. Tailored recommendations are incorporated immediately following the morning goal module.
- Affect + SAVOR: Participants receive affect-based goals for two weeks. In addition to the standard mHealth intervention, participants engage in the SAVOR enhancement to augment the treatment effects of the affect-based goals condition.
  Affect-Based Goals: On days participants plan to exercise, they engage in affect-based goal-setting sessions. Participants are asked to engage in a type or context of physical activity that allows them to experience positive affect.
  SAVOR Enhancement: The SAVOR enhancement will augment affect-based treatment effects by additionally implementing a brief savoring exercise on the smartphone during the evening goal session (after the self-monitoring module). Participants will respond to questions that are intended to enhance and prolong positive experiences during physical activity. To trigger attentional deployment, a common savoring strategy that involves intensifying experiences by focusing on them, participants will answer open-ended prompts. These prompts are drawn from a prompt pool with slightly varied wording to promote a sense of novelty.
- Affect + TYPE/CONTEXT + SAVOR: Participants receive affect-based goals for two weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT and SAVOR enhancements to augment the treatment effects of the affect-based goals condition.
  Affect-Based Goals: On days participants plan to exercise, they engage in affect-based goal-setting sessions. Participants are asked to engage in a type or context of physical activity that allows them to experience positive affect.
  TYPE/CONTEXT Enhancement: The TYPE/CONTEXT enhancement will augment affect-based treatment effects via tailored recommendations for activity types and contexts that satisfy personally important psychological needs as rated by each participant at baseline (see full description in previous groups)
  SAVOR Enhancement: The SAVOR enhancement will augment affect-based treatment effects by additionally implementing a brief savoring exercise on the smartphone during the evening goal session (after the self-monitoring module) (see full description in previous groups).
Period: Overall Study
Arm/Group | Intensity | Affect + TYPE/CONTEXT | Affect + SAVOR | Affect + TYPE/CONTEXT + SAVOR
Started | 9 | 10 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensity | Affect + TYPE/CONTEXT | Affect + SAVOR | Affect + TYPE/CONTEXT + SAVOR | Total
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.67 (9.042) | 46.30 (17.327) | 43.11 (13.004) | 51.56 (13.106) | 46.16 (13.422)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 6 | 20
  Male | 4 | 5 | 5 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 0 | 5
  Not Hispanic or Latino | 7 | 9 | 7 | 9 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 0 | 4
  White | 8 | 9 | 6 | 9 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.3942 (5.48859) | 35.0256 (5.72246) | 32.7438 (4.87365) | 32.7050 (5.36799) | 33.2660 (5.26874)
Household Income [Count of Participants; unit: Participants]
  Unsure | 0 | 0 | 2 | 1 | 3
  ≤ $44,999 | 1 | 2 | 1 | 3 | 7
  $45,000 to $84,999 | 2 | 2 | 2 | 3 | 9
  $85,000 to $124,999 | 1 | 4 | 1 | 2 | 8
  ≥ $125,000 | 5 | 2 | 3 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety Benchmark: Percentage of Participants Experiencing an Adverse Event
Description: An adverse event is that which is unexpected, related or possibly related to the study procedures, and serious (adversely affecting the balance of risks and benefits to participation, including incidents that require hospitalization, specialist treatment, or medical intervention). This refers to any adverse event that can be reasonably determined (at least in part) to be due to the study procedures and not due to a participant's underlying medical conditions or risk factor profile alone. This is assessed by official University of Southern California Institutional Review Board reporting procedures. The study's official "go/no-go" criterion is that less than 1% of participants experience an adverse event during the study.
Time Frame: Event onset reported as from first day of run-in period (i.e., day 1) to one week post-data collection (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | Intensity | Affect + TYPE/CONTEXT | Affect + SAVOR | Affect + TYPE/CONTEXT + SAVOR
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Reported adverse event | 0 | 0 | 0 | 0
  Did not report adverse event | 9 | 9 | 9 | 9

2. Primary Outcome: Efficacy Benchmark: Percentage of Participants With Increased Physical Activity Enjoyment
Description: During the exit interview, participants compare their experience with physical activity before and after participation in the eMOTION Study and are asked if they personally feel as if the degree of enjoyment they feel while engaging in physical activity changed or stayed the same. The percentage of participants responding affirmatively will be calculated. The "go/no-go criterion" is that ≥51% of participants in the affect-based conditions report a perceived increase in enjoyment of physical activity.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis explored whether participants who received affect-based goals (regardless of the specific TYPE/CONTEXT and/or SAVOR enhancements included) reported increased enjoyment. The three affect-based arms (affect + TYPE/CONTEXT [n=9], affect + SAVOR [n=9], affect + TYPE/CONTEXT + SAVOR [n=9]) were therefore considered to be a single collapsed sub-sample (n=27). This is because we did not have a large enough sample size to compare between the four groups.
Measure: Count of Participants; unit: Participants
Groups:
- Affect: Participants receive affect-based goals for two weeks. In addition to the standard mHealth intervention, participants engage in enhancements-- TYPE/CONTEXT, SAVOR, or both TYPE/CONTEXT and SAVOR-- to augment the treatment effects of the affect-based goals condition.
Arm/Group | Intensity | Affect
Number analyzed (Participants) | 9 | 27
Participants
  Enjoyment increased | 2 | 14
  Enjoyment stayed the same | 6 | 13
  Enjoyment decreased | 0 | 0
  Missing | 1 | 0

3. Primary Outcome: Accessibility/Usability Benchmark: System Usability Scale Score (0 to 100) for Daily Goal Sessions & Fitbit
Description: In the Post-Study Questionnaire, participants will rate the usability of the eMOTION Study's daily goal sessions and Fitbit Versa protocol via the System Usability Scale (SUS). The SUS has 10 items, and participants indicate their degree of agreement with each statement on a 5-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (5). The SUS is then scored by summing across items (all items are first rescored to a 0 to 4 scale, and even items are reverse-scored before summing) and then multiplying the sum by 2.5. The study's go/no-go criterion is that both the daily goal sessions and Fitbit protocols receive at least an average score (≥68) on the SUS.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: The study protocol and statistical analysis plan pre-specified that treatment arms would be assessed in a combined manner (i.e, as a full sample). This analysis explored the basic usability of the primary components (i.e., daily goal sessions, Fitbit Versa) used to deliver the eMOTION Study intervention, which were kept uniform for all participants, regardless of treatment arm (i.e., intensity-based goals, affect + TYPE/CONTEXT, affect + SAVOR, affect + TYPE/CONTEXT + SAVOR).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Full Sample: For the purposes of this outcome measure, all study participants-- regardless of their intensity/affect group-- are considered.
Arm/Group | Full Sample
Number analyzed (Participants) | 36
score on a scale
  Daily Goals Score | 72.4306 (17.21177)
  Fitbit Score | 73.0556 (22.85131)

4. Primary Outcome: Accessibility/Usability Benchmark: Percentage of Participants Rating Daily Goal Sessions and Fitbit Interface as Accessible
Description: The degree of accessibility of the daily goal sessions and fitbit interface for the study will also be assessed in the exit interview. Specifically, participants are asked a series of questions about whether they were able to read, understand, and select answers for Fitbit watch face surveys and use the exercise settings. They are also asked if they were able to red and understand the daily goal sessions on their phone. The go/no-go criterion is that at least 51% of participants respond affirmatively for each facet.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: The study protocol and statistical analysis plan pre-specified that treatment arms would be assessed in a combined manner (i.e, as a full sample). This analysis explored the basic accessibility/usability of the primary components (i.e., daily goal sessions, Fitbit Versa) used to deliver the eMOTION Study intervention, which were kept uniform for all participants, regardless of treatment arm (i.e., intensity-based goals, affect + TYPE/CONTEXT, affect + SAVOR, affect + TYPE/CONTEXT + SAVOR).
Measure: Count of Participants; unit: Participants
Arm/Group | Full Sample
Number analyzed (Participants) | 36
Participants
  Read Fitbit: No | 1
  Read Fitbit: Yes | 34
  Read Fitbit: Missing | 1
  Understand Fitbit: No | 3
  Understand Fitbit: Yes | 32
  Understand Fitbit: Missing | 1
  Select Fitbit answers: No | 2
  Select Fitbit answers: Yes | 33
  Select Fitbit answers: Missing | 1
  Use Fitbit exercise settings: No | 8
  Use Fitbit exercise settings: Yes | 27
  Use Fitbit exercise settings: Missing | 1
  Read daily goals: No | 1
  Read daily goals: Yes | 34
  Read daily goals: Missing | 1
  Understand daily goals: No | 1
  Understand daily goals: Yes | 34
  Understand daily goals: Missing | 1

5. Primary Outcome: Accessibility/Usability Benchmark: Physical Activity Recommendations Appropriately Consider Reported Constraints
Description: Participants are asked to indicate whether they have any constraints limiting their engagement in specific physical activity types or contexts as part of the baseline questionnaire. They also rate the relative importance of each of the psychological needs to them personally at baseline. For participants who receive the TYPE/CONTEXT enhancement with the affect-based goals, an algorithm produces physical activity recommendations based on their psychological needs that also considers their reported constraints. During the exit interview, participants in this group are asked whether they were able to follow the physical activity recommendations. The go/no-go criterion is that there is no pattern between the number of constraints reported at baseline and participants' reported ability to follow activity recommendations; therefore, we qualitatively compared the mean percentage of recommendations that participants could follow across constraint quartiles.
Time Frame: Assessed on date of baseline questionnaire completion and at 3 weeks (i.e., post-study)
Population: This analysis only applied to participants who received TYPE/CONTEXT recommendations. The two TYPE/CONTEXT arms (i.e., affect-based goals + TYPE/CONTEXT, affect-based goals + TYPE/CONTEXT + SAVOR) were combined and considered as a single sub-sample (N=18), since both received identical TYPE/CONTEXT treatment components. n=3 of these participants did not remember receiving TYPE/CONTEXT recommendations, so they were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage of recommendations
Groups:
- First Quartile (< 30.25 Constraints): Only participants who received the TYPE/CONTEXT enhancement (i.e., belonged to the affect-based goals + TYPE/CONTEXT or affect-based goals + TYPE/CONTEXT + SAVOR treatment arms) were included in the current analysis. Participants reported the number of activity types and contexts for which they had a constraint. The first quartile of total constraints-- or those who had the least number of constraints-- includes participants who reported having < 30.25 constrained activity types/contexts.
- Second Quartile (30.25 to < 37.00 Constraints): Only participants who received the TYPE/CONTEXT enhancement (i.e., belonged to the affect-based goals + TYPE/CONTEXT or affect-based goals + TYPE/CONTEXT + SAVOR treatment arms) were included in the current analysis. Participants reported the number of activity types and contexts for which they had a constraint. The second quartile of total constraints includes participants who reported having 30.25 to < 37.00 constrained activity types/contexts.
- Third Quartile (37.00 to < 41.75): Only participants who received the TYPE/CONTEXT enhancement (i.e., belonged to the affect-based goals + TYPE/CONTEXT or affect-based goals + TYPE/CONTEXT + SAVOR treatment arms) were included in the current analysis. Participants reported the number of activity types and contexts for which they had a constraint. The third quartile of total constraints includes participants who reported having 37.00 to <41.75 constrained activity types/contexts.
- Fourth Quartile (≥ 41.75 Constraints): Only participants who received the TYPE/CONTEXT enhancement (i.e., belonged to the affect-based goals + TYPE/CONTEXT or affect-based goals + TYPE/CONTEXT + SAVOR treatment arms) were included in the current analysis. Participants reported the number of activity types and contexts for which they had a constraint. The fourth quartile of total constraints-- or those with the most number of constraints-- includes participants who reported having ≥ 41.75 constrained activity types/contexts.
Arm/Group | First Quartile (< 30.25 Constraints) | Second Quartile (30.25 to < 37.00 Constraints) | Third Quartile (37.00 to < 41.75) | Fourth Quartile (≥ 41.75 Constraints)
Number analyzed (Participants) | 5 | 2 | 4 | 4
percentage of recommendations | 40 (54.8) | 50 (70.7) | 50 (57.7) | 25 (50.0)

6. Primary Outcome: Accessibility/Usability Benchmark: Percentage of Participants Rating Savoring Exercises as Accessible
Description: During the exit interview, participants who received the SAVOR enhancement with the affect-based goals will be asked whether they were generally able to understand and follow the savoring questions they received. The go/no-go criterion for accessibility is that ≥51% of participants reported being able to understand and follow the savoring questions.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis only applied to participants who received savoring exercises. The two SAVOR arms (i.e., affect-based goals + SAVOR, affect-based goals + TYPE/CONTEXT + SAVOR) were combined and considered as a single sub-sample (N=18), since both received identical SAVOR treatment components. n=4 of these participants did not remember receiving savoring exercises, so they were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- SAVOR Enhancement Sub-sample: Only participants who received the SAVOR enhancement (i.e., belonged to the affect-based goals + SAVOR or affect-based goals + TYPE/CONTEXT + SAVOR treatment arms) were included in the current analysis.
Arm/Group | SAVOR Enhancement Sub-sample
Number analyzed (Participants) | 14
Participants
  Understand savoring exercises: Yes | 12
  Understand savoring exercises: No | 2
  Follow savoring exercises: Yes | 12
  Follow savoring exercises: No | 2

7. Primary Outcome: Sustainability/Feasibility Benchmark: Fidelity of Auto-detection Algorithm
Description: Event-contingent surveys are triggered when Fitbit sensors detect physical activity via sufficiently-elevated 10-min rolling average heart rate (i.e., 55 to 60% of age-adjusted heart rate maximum). Using Fitabase data exports, the investigators will determine the percentage of correctly triggered surveys. The go/no-go criterion is that the auto-detection algorithm for physical activity correctly triggers event-contingent surveys ≥51% of the time.
Time Frame: From first full day of intervention (i.e., day 8) to last day of data collection (i.e., day 21)
Population: The study protocol and statistical analysis plan pre-specified that treatment arms would be assessed in a combined manner (i.e, as a full sample). The physical activity auto-detection algorithm was applied uniformly across all participants (N=36), regardless of treatment arm. The number of correctly-triggered surveys were divided by the total number of event-contingent surveys sent during the study (i.e., N=1555) in this analysis.
Measure: Count of Units; unit: Total event-contingent surveys
Units Other Than Participants: Total event-contingent surveys
Arm/Group | Full Sample
Number analyzed (Participants) | 36
Number analyzed (Total event-contingent surveys) | 1555
Total event-contingent surveys
  Surveys triggered successfully | 1555
  Surveys not triggered successfully | 0

8. Primary Outcome: Sustainability/Feasibility Benchmark: Research Staff Burden
Description: This benchmark determines if the level of burden for research staff is sustainable/feasible related to Fitbit technological and connectivity issues. Staff track Fitbit inventory and document technical difficulties that require a replacement device, as well as record all instances where they have to remind participants to sync the data in their Fitbit app due to > 48 h elapsing without data reaching Fitabase servers. Go/no-go criteria are that, over the course of the study, < 25% of participants need a replacement Fitbit due to technological issues and < 25% of participants are sent repeated (i.e., >1) reminders to sync their data.
Time Frame: From first day of run-in period (i.e., day 1) to last day of data collection (i.e., day 21)
Population: The study protocol and statistical analysis plan pre-specified that treatment arms would be assessed in a combined manner (i.e, as a full sample). This analysis focused on the basic sustainability/feasibility of Fitbit-related issues for study staff. Because all participants received Fitbit smartwatches that underwent uniform technological setup and connectivity procedures, each participant's treatment arm was irrelevant.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Sample
Number analyzed (Participants) | 36
Participants
  Replacement Fitbit required?: Yes | 0
  Replacement Fitbit required?: No | 36
  >1 reminders to sync data?: Yes | 0
  >1 reminders to sync data?: No | 36

9. Primary Outcome: Sustainability/Feasibility Benchmark: Satisfaction With Fitbit and Daily Goal Session Components
Description: The Delighted-Terrible Scale was used to assess how participants felt about the study's Fitbit and smartphone functions in the post-study questionnaire. Items asked how they felt about the Fitbit smartwatch exercise settings, notifications to complete surveys, and survey frequency and length (i.e., burden); as well as how they felt about the smartphone-based daily goal sessions and Fitbit app. Response options are: feeling delighted (7), pleased (6), mostly satisfied (5), mixed- about equally satisfied and dissatisfied (4), mostly dissatisfied (3), unhappy (2), terrible (1) -- OR -- neutral- neither satisfied nor dissatisfied (a), or never thought about it (b). The go/no-go criterion is that <70% of participants report feeling dissatisfied (considered to be a score of 1, 2, or 3) with any of the items.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: The study protocol and statistical analysis plan pre-specified that treatment arms would be assessed in a combined manner (i.e, as a full sample). All participants engaged with the most basic Fitbit and smartphone-based components in the same way, regardless of their treatment arms. All items asked about study elements that were kept uniform across participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Sample
Number analyzed (Participants) | 36
Participants
  Exercise settings: Satisfied | 30
  Exercise settings: Dissatisfied | 6
  Exercise settings: Missing | 0
  Survey notifications: Satisfied | 24
  Survey notifications: Dissatisfied | 12
  Survey notifications: Missing | 0
  Survey burden: Satisfied | 22
  Survey burden: Dissatisfied | 14
  Survey burden: Missing | 0
  Daily goal sessions: Satisfied | 31
  Daily goal sessions: Dissatisfied | 3
  Daily goal sessions: Missing | 2
  Fitbit app: Satisfied | 33
  Fitbit app: Dissatisfied | 3
  Fitbit app: Missing | 0

10. Primary Outcome: Sustainability/Feasibility Benchmark: Dissatisfaction With TYPE/CONTEXT Recommendations
Description: During the post-study questionnaire, participants who received recommendations for the specific types or contexts of physical activity to do (i.e., were in the affect-based goals + TYPE/CONTEXT or affect-based goals + TYPE/CONTEXT + SAVOR groups) will complete the Delighted-Terrible Scale. They are asked how they felt about the physical activity type/context recommendations they received. Response options are feeling delighted (7), pleased (6), mostly satisfied (5), mixed- about equally satisfied and dissatisfied (4), mostly dissatisfied (3), unhappy (2), terrible (1) -- OR -- neutral- neither satisfied nor dissatisfied (a), or never thought about it (b). The go/no-go criterion is that <70% of participants report feeling dissatisfied (score of 1 to 3) with physical activity recommendations.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis only applied to participants who received TYPE/CONTEXT recommendations. The two TYPE/CONTEXT arms (i.e., affect-based goals + TYPE/CONTEXT, affect-based goals + TYPE/CONTEXT + SAVOR) were combined and considered as a single sub-sample (N=18), since both received identical TYPE/CONTEXT treatment components. Of these participants, n=3 did not remember receiving TYPE/CONTEXT recommendations, and an additional n=2 failed to respond, so they were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- TYPE/CONTEXT Enhancement Sub-sample: Only participants who received the TYPE/CONTEXT enhancement (i.e., belonged to the affect-based goals + TYPE/CONTEXT or affect-based goals + TYPE/CONTEXT + SAVOR treatment arms) were included in the current analysis.
Arm/Group | TYPE/CONTEXT Enhancement Sub-sample
Number analyzed (Participants) | 13
Participants
  Satisfied | 10
  Dissatisfied | 3

11. Primary Outcome: Sustainability/Feasibility Benchmark: Dissatisfaction With SAVOR Questions
Description: During the post-study questionnaire, participants in the affect-based goals + SAVOR or affect-based goals + TYPE/CONTEXT + SAVOR groups will complete the validated Delighted-Terrible Scale. They are asked how they felt about the savoring questions they received. Response options are: feeling delighted (7), pleased (6), mostly satisfied (5), mixed- about equally satisfied and dissatisfied (4), mostly dissatisfied (3), unhappy (2), terrible (1) -- OR -- neutral- neither satisfied nor dissatisfied (a), or never thought about it (b). The go/no-go criterion is that <70% of participants report feeling dissatisfied (score of 1 to 3) with savoring questions.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis only applied to participants who received SAVOR questions. The two SAVOR arms (i.e., affect-based goals + SAVOR, affect-based goals + TYPE/CONTEXT + SAVOR) were combined and considered as a single sub-sample (N=18), since both received identical SAVOR treatment components. Of these participants, n=4 did not remember receiving TYPE/CONTEXT recommendations, and an additional n=2 did not respond, so they were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SAVOR Enhancement Sub-sample
Number analyzed (Participants) | 12
Participants
  Satisfied | 12
  Dissatisfied | 0

12. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal for Males vs. Females
Description: Equity was explored based on whether accessibility/usability were approximately the same between males vs. females. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to sex-at-birth (male vs. female), regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample (N=36) were split into two sub-groups based on sex.
Measure: Count of Participants; unit: Participants
Groups:
- Male: Participants who reported their sex at birth as male were included in this group.
- Female: Participants who reported their sex at birth as female were included in this group.
Arm/Group | Male | Female
Number analyzed (Participants) | 17 | 19
Participants
  Daily Goal Session: Accessible/usable | 11 | 12
  Daily Goal Session: Not accessible/usable | 6 | 7
  Fitbit Protocol: Accessible/usable | 13 | 13
  Fitbit Protocol: Not accessible/usable | 4 | 6

13. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal for Males vs. Females
Description: Equity was explored based on whether efficacy was approximately the same between males vs. females. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 17 | 19
Participants
  Efficacious | 6 | 10
  Not Efficacious | 11 | 8
  Missing | 0 | 1

14. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal for White vs. Non-white Participants
Description: Equity was explored based on whether accessibility/usability was approximately the same between white vs. non-white participants. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to race (white vs. non-white), regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample were split into two sub-groups based on race.
Measure: Count of Participants; unit: Participants
Groups:
- White: Participants who reported their race as white were included in this group.
- Non-white: Participants who reported their race as anything other than white were included in this group.
Arm/Group | White | Non-white
Number analyzed (Participants) | 31 | 5
Participants
  Daily goal sessions: Accessible/usable | 19 | 4
  Daily goal sessions: Not accessible/usable | 12 | 1
  Fitbit protocol: Accessible/usable | 21 | 5
  Fitbit protocol: Not accessible/usable | 10 | 0

15. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal for White vs. Non-white Participants
Description: Equity was explored based on whether efficacy was approximately the same between white vs. non-white participants. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | White | Non-white
Number analyzed (Participants) | 31 | 5
Participants
  Efficacious | 12 | 4
  Not efficacious | 18 | 1
  Missing | 1 | 0

16. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal for Hispanic vs. Non-Hispanic Participants
Description: Equity was explored based on whether accessibility/usability was approximately the same between Hispanic vs. non-Hispanic participants. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to ethnicity (Hispanic vs. non-Hispanic), regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample were split into two sub-groups based on ethnicity.
Measure: Count of Participants; unit: Participants
Groups:
- Hispanic: Participants who reported their ethnicity as Hispanic were included in this group.
- Non-Hispanic: Participants who reported their ethnicity as non-Hispanic were included in this group.
Arm/Group | Hispanic | Non-Hispanic
Number analyzed (Participants) | 4 | 32
Participants
  Daily goal sessions: Accessible/usable | 2 | 21
  Daily goal sessions: Not accessible/usable | 2 | 11
  Fitbit protocol: Accessible/usable | 2 | 24
  Fitbit protocol: Not accessible/usable | 2 | 8

17. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal for Hispanic vs. Non-Hispanic Participants
Description: Equity was explored based on whether efficacy was approximately the same between Hispanic vs. non-Hispanic participants. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Hispanic | Non-Hispanic
Number analyzed (Participants) | 4 | 32
Participants
  Efficacious | 1 | 15
  Not efficacious | 3 | 16
  Missing | 0 | 1

18. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal Across Income Categories
Description: Equity was explored based on whether accessibility/usability was approximately the same between various income categories. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to annual income, regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample were split into five sub-groups based on income.
Measure: Count of Participants; unit: Participants
Groups:
- Unsure of Income: Participants who were unsure of their annual income were included in this group.
- ≤ $44,999: Participants who reported their annual income as ≤ $44,999 were included in this group.
- $45,000 to $84,999: Participants who reported their annual income as $45,000 to $84,999 were included in this group.
- $85,000 to $124,999: Participants who reported their annual income as $85,000 to $124,999 were included in this group.
- ≥ $125,000: Participants who reported their annual income as ≥ $125,000 were included in this group.
Arm/Group | Unsure of Income | ≤ $44,999 | $45,000 to $84,999 | $85,000 to $124,999 | ≥ $125,000
Number analyzed (Participants) | 3 | 6 | 9 | 8 | 10
Participants
  Daily goal sessions: Accessible/usable | 1 | 3 | 6 | 4 | 9
  Daily goal sessions: Not accessible/usable | 2 | 3 | 3 | 4 | 1
  Fitbit protocol: Accessible/usable | 3 | 3 | 6 | 5 | 9
  Fitbit protocol: Not accessible/usable | 0 | 3 | 3 | 3 | 1

19. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal Across Income Categories
Description: Equity was explored based on whether efficacy was approximately the same between various income categories. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Unsure of Income | ≤ $44,999 | $45,000 to $84,999 | $85,000 to $124,999 | ≥ $125,000
Number analyzed (Participants) | 3 | 6 | 9 | 8 | 10
Participants
  Efficacious | 0 | 1 | 8 | 3 | 4
  Not efficacious | 3 | 5 | 1 | 5 | 5
  Missing | 0 | 0 | 0 | 0 | 1

20. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal Across Age Categories
Description: Equity was explored based on whether accessibility/usability was approximately the same between age quartiles. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to age, regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample were split into four quartiles based on age.
Measure: Count of Participants; unit: Participants
Groups:
- ≤ 37 Years: Participants who reported their age as ≤ 37 years were included in this group.
- 38 to 43 Years: Participants who reported their age as 38 to 43 years were included in this group.
- 44 to 58 Years: Participants who reported their age as 44 to 58 years were included in this group.
- ≥ 59 Years: Participants who reported their age as ≥ 59 years were included in this group.
Arm/Group | ≤ 37 Years | 38 to 43 Years | 44 to 58 Years | ≥ 59 Years
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Daily goal sessions: Accessible/usable | 3 | 6 | 8 | 6
  Daily goal sessions: Not accessible/usable | 6 | 3 | 1 | 3
  Fitbit protocol: Accessible/usable | 6 | 6 | 8 | 6
  Fitbit protocol: Not accessible/usable | 3 | 3 | 1 | 3

21. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal Across Age Categories
Description: Equity was explored based on whether efficacy was approximately the same between age quartiles. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | ≤ 37 Years | 38 to 43 Years | 44 to 58 Years | ≥ 59 Years
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Efficacious | 5 | 2 | 4 | 5
  Not efficacious | 4 | 7 | 4 | 4
  Missing | 0 | 0 | 1 | 0

22. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal for Participants With Overweight vs. Obesity
Description: Equity was explored based on whether accessibility/usability was approximately the same between participants with overweight vs. obesity. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to BMI status (overweight vs. obese), regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample were split into two sub-groups based on BMI status.
Measure: Count of Participants; unit: Participants
Groups:
- Overweight: Participants reported their height and weight. BMI was then calculated as kg/m^2. Participants with a BMI of 25 to 29.9 were categorized as overweight.
- Obese: Participants reported their height and weight. BMI was then calculated as kg/m^2. Participants with a BMI ≥ 30.0 were categorized as obese.
Arm/Group | Overweight | Obese
Number analyzed (Participants) | 12 | 24
Participants
  Daily goal sessions: Accessible/usable | 8 | 15
  Daily goal sessions: Not accessible/usable | 4 | 9
  Fitbit protocol: Accessible/usable | 10 | 16
  Fitbit protocol: Not accessible/usable | 2 | 8

23. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal for Participants With Overweight vs. Obesity
Description: Equity was explored based on whether efficacy was approximately the same between participants with overweight vs. obesity. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Overweight | Obese
Number analyzed (Participants) | 12 | 24
Participants
  Efficacious | 5 | 11
  Not efficacious | 6 | 13
  Missing | 1 | 0

24. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal Across Mobility Categories
Description: Equity was explored based on whether accessibility/usability was approximately the same between mobility quartiles. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to mobility, regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample were split into four quartiles based on mobility.
Measure: Count of Participants; unit: Participants
Groups:
- First Quartile (Mobility Score ≤ 13.5): Participants rated the degree to which they had agreed with each of five mobility-related statements using a 10-point sliding scale (with markers "Not at all true" [1], "Moderately true" [5], "Completely true" [10]). The total mobility score was then tallied across items, with lower total scores signifying the least trouble with mobility and higher total scores signifying the most trouble with mobility. Participants in the lowest quartile (i.e., with the least mobility trouble; mobility scores ≤ 13.5) were included in this group.
- Second Quartile (Mobility Score 13.6 to 18.5): Participants rated the degree to which they had agreed with each of five mobility-related statements using a 10-point sliding scale (with markers "Not at all true" [1], "Moderately true" [5], "Completely true" [10]). The total mobility score was then tallied across items, with lower total scores signifying the least trouble with mobility and higher total scores signifying the most trouble with mobility. Participants in the second-lowest quartile (i.e., mobility scores 13.6 to 18.5) were included in this group.
- Third Quartile (Mobility Score 18.6 to 28.5): Participants rated the degree to which they had agreed with each of five mobility-related statements using a 10-point sliding scale (with markers "Not at all true" [1], "Moderately true" [5], "Completely true" [10]). The total mobility score was then tallied across items, with lower total scores signifying the least trouble with mobility and higher total scores signifying the most trouble with mobility. Participants in the second-highest quartile (i.e., mobility scores 18.6 to 28.5) were included in this group.
- Fourth Quartile (Mobility Score ≥ 28.6): Participants rated the degree to which they had agreed with each of five mobility-related statements using a 10-point sliding scale (with markers "Not at all true" [1], "Moderately true" [5], "Completely true" [10]). The total mobility score was then tallied across items, with lower total scores signifying the least trouble with mobility and higher total scores signifying the most trouble with mobility. Participants in the highest quartile (i.e., with the most mobility trouble; mobility scores ≥ 28.6) were included in this group.
Arm/Group | First Quartile (Mobility Score ≤ 13.5) | Second Quartile (Mobility Score 13.6 to 18.5) | Third Quartile (Mobility Score 18.6 to 28.5) | Fourth Quartile (Mobility Score ≥ 28.6)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Daily goal sessions: Accessible/usable | 6 | 6 | 6 | 5
  Daily goal sessions: Not accessible/usable | 3 | 3 | 3 | 4
  Fitbit protocol: Accessible/usable | 7 | 8 | 7 | 4
  Fitbit protocol: Not accessible/usable | 2 | 1 | 2 | 5

25. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal Across Mobility Categories
Description: Equity was explored based on whether efficacy was approximately the same between mobility quartiles. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | First Quartile (Mobility Score ≤ 13.5) | Second Quartile (Mobility Score 13.6 to 18.5) | Third Quartile (Mobility Score 18.6 to 28.5) | Fourth Quartile (Mobility Score ≥ 28.6)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Efficacious | 5 | 4 | 5 | 2
  Not efficacious | 3 | 5 | 4 | 7
  Missing | 1 | 0 | 0 | 0

26. Primary Outcome: Equity Benchmark: Accessibility/Usability Approximately Equal Across Physical Constraint Categories
Description: Equity was explored based on whether accessibility/usability was approximately the same between physical constraint tertiles. The percentage of participants who rated the daily goal sessions and Fitbit protocol as sufficiently accessible/usable (i.e., scored the daily goal sessions and Fitbit protocol at-or-above the System Usability Scale's validated cutoff of 68) were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: This analysis was concerned with the basic equity of the eMOTION Study intervention related to physical constraints, regardless of the specific treatment arm that participants were in. Therefore, participants from the full sample were split into three tertiles based on physical constraints.
Measure: Count of Participants; unit: Participants
Groups:
- First Tertile (no Constraints): For 47 types of physical activities, participants indicated whether they were physically able or unable to perform each one. The number of activities they were physically unable to perform was summed to create a total constraint score (ranging from 0 [no physical constraints] to 47 [maximum physical constraints]). Participants in the first tertile (i.e., no constraints reported) were included in this group.
- Second Tertile (1 to 4 Constraints): For 47 types of physical activities, participants indicated whether they were physically able or unable to perform each one. The number of activities they were physically unable to perform was summed to create a total constraint score (ranging from 0 [no physical constraints] to 47 [maximum physical constraints]). Participants in the second tertile (i.e., 1 to 4 constraints reported) were included in this group.
- Third Tertile (≥ 5 Constraints): For 47 types of physical activities, participants indicated whether they were physically able or unable to perform each one. The number of activities they were physically unable to perform was summed to create a total constraint score (ranging from 0 [no physical constraints] to 47 [maximum physical constraints]). Participants in the third tertile (i.e., ≥ 5 constraints reported) were included in this group.
Arm/Group | First Tertile (no Constraints) | Second Tertile (1 to 4 Constraints) | Third Tertile (≥ 5 Constraints)
Number analyzed (Participants) | 15 | 12 | 9
Participants
  Daily goal sessions: Accessible/usable | 10 | 9 | 4
  Daily goal sessions: Not accessible/usable | 5 | 3 | 5
  Fitbit protocol: Accessible/usable | 12 | 9 | 5
  Fitbit protocol: Not accessible/usable | 3 | 3 | 4

27. Primary Outcome: Equity Benchmark: Efficacy Approximately Equal Across Physical Constraint Categories
Description: Equity was explored based on whether efficacy was approximately the same between physical constraint categories. The percentage of participants who reported experiencing (i.e., efficacious) or not experiencing (i.e., not efficacious) an increase in enjoyment for physical activity during the study were calculated.
Time Frame: Reported at 3 weeks (i.e., post-study)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | First Tertile (no Constraints) | Second Tertile (1 to 4 Constraints) | Third Tertile (≥ 5 Constraints)
Number analyzed (Participants) | 15 | 12 | 9
Participants
  Efficacious | 6 | 7 | 3
  Not efficacious | 8 | 5 | 6
  Missing | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks (from first day of run-in period [i.e., day 1] to one week post-data collection [week 4])
Arm/Group | Intensity | Affect + TYPE/CONTEXT | Affect + SAVOR | Affect + TYPE/CONTEXT + SAVOR
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT06125964/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT06125964/ICF_001.pdf